CLINICAL TRIAL: NCT00369200
Title: A Phase 1 Study of AFP464 (Aminoflavone Prodrug) in Patients With Advanced Solid Tumors
Brief Title: AFP464 in Treating Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00163; NCI-2009-00163 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000492006; 2006-011 (Other: Wayne State University); 7378 (Other: CTEP); U01CA062487 (NIH)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific

ARMS (1):
- Arm I (Experimental): Patients receive AFP464 IV over 3 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.
  Cohorts of 2-6 patients receive escalating doses of AFP464 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which ≤ 1 of 6 patients experience dose-limiting toxicity. An additional 10 patients whose tumor is amenable to biopsy are treated at the MTD.
  Patients undergo blood collection periodically for pharmacokinetic and pharmacodynamic studies. Patients treated at the MTD also undergo tumor tissue biopsies periodically for additional pharmacodynamic and correlative biomarker studies.
  After completion of study treatment, patients are followed for 4 weeks.
  Interventions: Drug: AFP464; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: AFP464 — Given IV
Other: laboratory biomarker analysis — Correlative study
Other: pharmacological study — Correlative study
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of AFP464 in treating patients with advanced solid tumors. Drugs used in chemotherapy, such as AFP464, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose-limiting toxicity and maximum tolerated dose of AFP464 in patients with advanced solid tumors.

II. Assess the safety and tolerability of this drug in these patients.

SECONDARY OBJECTIVES:

I. Observe clinical response in patients treated with this drug. II. Characterize the pharmacokinetics of this drug in these patients. III. Determine the clinical significance of genetic polymorphisms on the genes coding metabolizing enzymes (e.g., CYP1A1, 1A2, 2C9, 2C19, and SULTA1) and on the disposition and efficacy/toxicity of AFP464 and AF.

OUTLINE: This a dose-escalation, multicenter study.

Patients receive AFP464 IV over 3 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.

Cohorts of 2-6 patients receive escalating doses of AFP464 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which ≤ 1 of 6 patients experience dose-limiting toxicity. An additional 10 patients whose tumor is amenable to biopsy are treated at the MTD.

Patients undergo blood collection periodically for pharmacokinetic and pharmacodynamic studies. Patients treated at the MTD also undergo tumor tissue biopsies periodically for additional pharmacodynamic and correlative biomarker studies.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Bilirubin normal
* Platelet count >= 100,000/mm³
* AST and ALT =< 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance >= 60 mL/min
* Adequate pulmonary function
* DLCO =< grade 1
* No symptomatic pulmonary disease
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Negative pregnancy test
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to AFP464
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit study compliance
* No smoking within the past 30 days; must be willing and able to completely refrain from smoking during study participation
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin C, or bleomycin) and recovered
* At least 4 weeks since prior radiotherapy; no prior thoracic radiotherapy; no prior radiotherapy to >= 50% of total marrow volume
* More than 4 weeks since prior experimental therapy (non-FDA-approved agents), immunotherapy, or targeted agents and recovered
* More than 8 weeks since prior UCN-01
* More than 2 weeks since prior hormonal therapy except for patients on androgen suppression for prostate cancer
* Concurrent androgen suppression allowed in patients with prostate cancer
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* Histologically confirmed malignant solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Tumor amenable to biopsy (maximum tolerated dose expansion cohort)
* No known brain metastases
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* Absolute neutrophil count >= 1,500/mm³
* No other concurrent anticancer agents or therapies
* Renal cell cancer, breast cancer, and non-small cell lung cancer encouraged

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-06; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose determined by dose-limiting toxicity | 28 days
Types and grades of toxicity | Up to 4 weeks
  Full frequency distributions of grade of toxicity, by toxicity type, will be generated, by dose level. Among all treated patients, both point and exact confidence interval estimates of the rate of every specific type of Grade 3-4 toxicity will be calculated, by dose level. Grade 2 DLCO rates (point and confidence level) will also be computed, by dose level.

SECONDARY OUTCOMES:
Pharmacokinetic, pharmacodynamic, and pharmacogenomic parameters | Up to 4 weeks
Response rate | Up to 4 weeks
  Point and exact confidence interval estimates of response rate will be provided for all eligible patients combined, and if warranted, by specific dose levels.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia LoRusso, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States